CLINICAL TRIAL: NCT06972693
Title: Evaluating the Feasibility of NGS-based Germline and Somatic Genetic Testing in Ovarian Carcinoma. The PERSONA-ovary Trial
Brief Title: NGS-based Germline and Somatic Genetic Test in Ovarian Carcinoma
Acronym: PERSONA-Ovary
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 791
Record Dates: First submitted 2025-01-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Intervention Model Description: prospective observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRCA testing (Other)
  Interventions: Genetic: BRCA testing

INTERVENTIONS:
Genetic: BRCA testing — BRCA 1 and 2 testing

SUMMARY:
For patients with ovarian cancer and biologically related diseases, the implementation of genetic testing in the decision-making process could have an impact both on the risk management for the patient and his/her family, but also, more importantly, on the therapeutic management.

The identification of genetically predisposed subjects can suggest risk reduction strategies that may involve bilateral salpingo-oophorectomy, mastectomy or long-term medical approaches. In the advanced setting, genetic testing may influence the decision for medical therapy (e.g. use of platinum derivatives or PARP inhibitors in patients with "BRCAness+" ovarian cancer).

The selection of patients for genetic testing has so far been restricted to patients with a strong family history of breast and ovarian cancer. It is now clear that the strict application of this criterion will result in a substantial number of people with a missed BRCA mutation.

Systematic large-scale genetic testing, simultaneously on germline and somatic tissues, is likely to improve decision-making algorithms in ovarian cancer patients. The feasibility of such an approach in the clinical setting, in terms of response times compatible with clinical needs and sensitivity comparable if not superior to single-gene tests, needs to be demonstrated before such diagnostic platforms can be routinely implemented in the diagnostic workflow.

This is the aim of the present study.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or higher
2. has signed informed consent
3. histologically confirmed ovarian cancer, Fallopian tube cancer, or primary peritoneal cancer.
4. Any stage is admitted
5. Any histology is admitted
6. availability of surgical/bioptic material. Formalin-fixed, paraffinembedded or frozen specimens are both allowed, with no time limitation

Exclusion Criteria:

1. unable or unwilling to receive genetic counseling

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of clinically relevant mutations in ovarian cancer riskassociated genes | 3 months
  evaluate prevalence of clinically relevant mutations in ovarian cancer risk associated genes
Percentage of informative specimens | 3 months
  Percentage of informative specimens
Genetic test turnaround time | 3 months
  Evaluate Genetic test turnaround time

SECONDARY OUTCOMES:
Incidence of all other mutations | 3 months
  Incidence of all other mutations
progression-free survival | 10 years
  progression-free survival
overall survival | 10 years
  overall survival
Comparison of mutational profile across platforms: Devyser vs GerSom for BRC1/BRCA2 | 3 months
  Comparison of mutation in BRC1/BRCA2 genes between Devyser vs GerSom platform
Comparison of mutational profile across platforms: Trusight vs GerSom for all variants covered by both panels | 3 months
  Comparison of all gene mutations between Trusight and GerSom platform

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No